CLINICAL TRIAL: NCT02788305
Title: Effect of Maternal Obesity on Labour Induction in Postdate Pregnancy
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, heba mahmoud ibrahim marie, lecturer at kaselaini hospitals, Kasr El Aini Hospital
Other Study IDs: 9898
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Induced; Birth
MeSH Terms: conditions — Obesity | interventions — Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non obese: BMI<30. Misoprostol is given for induction of labour according to Bishop score
  Interventions: Drug: Misoprostol
- obese: BMI>30. Misoprostol is given for induction of labour according to Bishop score
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Misoprostol 25 micrograms every 6 hours will be given to obese and non obese groups

SUMMARY:
This study investigate the progression of labour in 144 normal weight pregnant women (BMI <30) and 144 obese pregnant women (BMI >30) , not in labor admitted for induction of labor. These women are to be investigated for success of induction of labor.

DETAILED DESCRIPTION:
* This prospective study will be conducted for 144 obese and 144 non obese ), post date (>41 wks), not in labor.
* Woman is classified as obese if BMI >=30.
* Prolonged pregnancy was defined as delivery on or after (41+0 weeks) of gestation.
* First informed consent will be obtained.
* Determination of gestational age
* Proper history taking, general and abdominal examinations will be done then digital examination will be performed to determine bishop score.
* And obstetric U/S scan will be done and by which the following data will be obtained :

  * Fetal biometry
  * Fetal heart activity
  * Presentation
  * Localization of the placenta.
  * Amount of amniotic fluid.
  * Exclude multifetal pregnancy.
* Induction of labor will be done using vaginal misoprostol according to the estimated Bishop score.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman.

  * Post date >= 41 weeks.
  * Absent onset of labor.
  * Patient acceptance to join the study after signing an informed consent.

Exclusion Criteria:

* Placenta previa and or vasa previa.
* Previous caesarean section(CS).
* Multiple gestation
* Any patient who will refuse to be a part of the study.
* Intra- uterine fetal death (IUFD).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 144 pregnant women with BMI >= 30 and 144 pregnant women with BMI <30, post date >= 41 wks, not in labor admitted in Kaselaini H for induction of labor.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
route of delivery vaginal or caesarean section. | 48 hours from the start of induction
  Partogram is used to access the progress of labour

SECONDARY OUTCOMES:
maternal haemorrhage | 48 hours from the start of induction
  Calculating number of soaked pads

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Marie, M.D., Principal Investigator — KasrElaini Hospital
Locations (1):
- Kasr wl aini hospitals, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, El-Semary AM, Marie HM, Belal DS, Hany A, Taymour MA, Omran EF, Elbaradie SMY, Mohamed MAK. Effect of maternal obesity on labor induction in postdate pregnancy. Arch Gynecol Obstet. 2018 Jul;298(1):45-50. doi: 10.1007/s00404-018-4767-8. Epub 2018 Apr 2. PMID 29610945